CLINICAL TRIAL: NCT01204450
Title: A Multi-center Phase I Trial of Temsirolimus in Combination With Valproic Acid in Children and Adolescents With Multiply Relapsed Pediatric Solid Tumors
Brief Title: Temsirolimus and Valproic Acid in Treating Young Patients With Relapsed Neuroblastoma, Bone Sarcoma, or Soft Tissue Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding has become unavailable
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0901; P30CA016086 (NIH); CDR0000665319 (Other: PDQ)
Record Dates: First submitted 2010-09-16; First posted 2010-09-17 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Brain and Central Nervous System Tumors; Neuroblastoma; Sarcoma; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: recurrent childhood brain tumor; recurrent childhood rhabdomyosarcoma; recurrent childhood soft tissue sarcoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent neuroblastoma; recurrent osteosarcoma; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Central Nervous System Neoplasms; Neuroblastoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Osteosarcoma | interventions — temsirolimus; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Temsirolimus + Valproic Acid (Other): Drug: temsirolimus 60-230mg/m2 weekly during each 28 day course, for up to 12 courses
  Drug: valproic acid (VPA) All patients will be given oral VPA (5 mg/kg, 3 times a day for each 28 day course, up to 12 courses
  Interventions: Drug: Temsirolimus; Drug: Valproic Acid

INTERVENTIONS:
Drug: Temsirolimus — 60-230mg/m2 weekly during each 28 day course, for up to 12 courses
  Other Names: Torisel
Drug: Valproic Acid — All patients will be given oral VPA (5 mg/kg, 3 times a day for each 28 day course, up to 12 courses
  Other Names: VPA

SUMMARY:
RATIONALE: Drugs such as temsirolimus and valproic acid may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Valproic acid may also stop the growth of solid tumors by blocking blood flow to the tumor.

PURPOSE: This phase I trial is studying the side effects and the best dose of temsirolimus when given together with valproic acid in treating young patients with relapsed neuroblastoma, bone sarcoma, or soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify the maximum-tolerated dose of temsirolimus in combination with valproic acid in highly pretreated pediatric patients with refractory solid tumors.

Secondary

* To estimate the objective response rate in patients treated with this regimen.
* To estimate the progression-free survival of patients treated with this regimen.
* To explore the association between tumor IGF-IR, mTOR expression, HDAC, autophagy biomarkers, and sera levels of temsirolimus, valproate, and VEGF-A with toxicity and disease response.
* To evaluate the ability of selected member divisions of a newly developed North Carolina-based pediatric oncology consortium to cooperate in clinical trials.

OUTLINE: This a multicenter, dose-escalation study of temsirolimus.

Patients receive temsirolimus IV over 30-60 minutes on days 1, 8, 15, and 22 and oral valproic acid* 3 times daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study for pharmacokinetic and VEGF-A studies. Tumor tissue samples from archived biopsy are also analyzed for IGF-IR, mTOR expression, HDAC, and autophagy biomarkers.

After completion of study therapy, patients are followed every 3 months for 1 year, every 4 months for 2 years, and then every 6 months for 2 years.

NOTE: * Doses of valproic acid are titrated beginning 3-7 days prior to starting temsirolimus to achieve plasma levels of 75-100 µg/mL.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor at original diagnosis, including the following:

  * Neuroblastoma
  * Bone sarcomas (primary neuroectodermal tumors/ Ewing sarcoma (PNET/ES), osteosarcoma)
  * Soft tissue sarcomas (rhabdosarcoma and related tumors)
* Histologically confirmed of relapsed disease is highly recommended but not mandatory
* Measurable disease according to RECIST
* Refractory or progressive disease after ≥ 1 and ≤ 4 prior chemotherapy regimens

  * Patients with neuroblastoma, PNET/ES, or rhabdosarcoma must have failed a cyclophosphamide/topotecan-containing regimen
  * Stem cell transplantation, including preparative regimen and post-transplant immunotherapy, is considered to be 1 regimen

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (or Lansky PS 50-100%)
* Life expectancy ≥ 8 weeks
* ANC ≥ 750/mm^3
* Platelet count ≥ 75,000/mm^3 (transfusion independent)
* Hemoglobin 8.0 g/dL (may receive RBC transfusions)

  * Patients with tumor metastatic to bone marrow are allowed to receive transfusions to maintain hemoglobin and platelet counts
* Serum creatinine normal
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN) OR direct bilirubin < 1.0 mg/dL (if total bilirubin > 2.0 mg/dL)
* ALT < 5 times ULN
* Negative pregnancy test
* Not pregnant or nursing
* Fertile patients must use effective contraception
* Families must be able to give consent in English or Spanish
* No allergy to H1 antihistamines

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior chemotherapy, immunotherapy, or radiotherapy and recovered
* No concurrent anticonvulsants, including valproic acid
* No concurrent strong inducers or inhibitors of CYP3A4, including grapefruit juice

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of temsirolimus in combination with valproic acid | 4 weeks
  The planned starting dose of Temsirolimus is 60mg/M2. The traditional 3+3 design will be used, where the MTD is defined as the dose with the probability of a DLT of 0.20

SECONDARY OUTCOMES:
Objective response rate | every 12 weeks
  Each patient will be classified according to their "best response". Best response is determined from the sequence of the objective statuses as described in RECIST 1.1
Progression-free survival | 3 years
  If the patient's disease has not progressed at the time protocol-directed therapy is complete, any tumor assessments available during the follow-up period (up to 3 years) will be evaluated using RECSIT 1.1
Temsirolimus pharmakokinetic parameters (Maximum plasma concentration) | doses 1 and 5
  Blood will be drawn prior to, 30 minutes, 1hr, 2hr, 5hr, 24hr after completion of doses 1 and 5. Levels of Temsirolimus will be measured using validated liquid chromatography and tandem mass spectroscopic methods

CONTACTS AND LOCATIONS:
Overall Officials: Julie Blatt, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Carolina Healthcare System, Charlotte, North Carolina